CLINICAL TRIAL: NCT02703493
Title: A Phase I Trial of IMRT With Dose-Escalated Image-Guided Stereotactic Radiosurgery (SRS) Boost for Human Papilloma Virus (HPV)- Unassociated Oropharyngeal Cancer
Brief Title: Image-Guided Stereotactic Radiosurgery (SRS) Boost for HPV-Oropharyngeal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Maged Ghaly, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-309A
Record Dates: First submitted 2015-12-15; First posted 2016-03-09 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cancer of the Oropharynx
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Dose escalation of radiation therapy for high risk oropharyngeal cancer
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cohort 1 (Experimental): Patients will receive 6 weeks of Intensity-Modulated Radiation Therapy (IMRT) (standard of care) followed by the dose escalated stereotactic radiosurgery (SRS Boost). Cohort 1 will receive 8 Gy in a single fraction, cohort 2 will receive 10 Gy in a single fraction and cohort 3 will receive 10 Gy split into two fractions.
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Patients will receive 6 weeks of IMRT (standard of care) followed by the stereotactic radiosurgery (SRS Boost). Dose of the boost is reliant on which cohort the patient is assigned to. Cohort 1 will receive 8 Gy, Cohort 2 will receive 10 Gy in a single fraction, Cohort 3 will receive 10 Gy split into two fractions.
  Other Names: SRS

SUMMARY:
This is a Phase I study looking to evaluate the safety of dose escalated stereotactic radiotherapy (SRS) without exceeding the maximum tolerated dose in patients with high-risk human papilloma virus (HPV)- unassociated oropharyngeal squamous cancer.

DETAILED DESCRIPTION:
Human Papilloma Virus (HPV) is frequently found within tumor cells removed from patients diagnosed with oropharynx cancer. Tumors which do not contain HPV virus (termed "HPV-Negative") are not cured as frequently by radiation therapy. Tumors which do contain HPV in patients who have a history of cigarette smoking also are not cured as frequently by radiation.

One way to potentially overcome this challenge is to deliver a more intense dose of radiation treatment to the tumor. The standard way to deliver radiation, termed Intensity Modulated Radiotherapy (IMRT), can protect normal tissues near tumors to a certain degree but not completely. Stereotactic radiosurgery (SRS) is a technique which can deliver radiation more precisely.

This trial will test the safety of treating HPV-unassociated oropharynx tumors to higher radiation doses wth SRS (termed a "boost") after a standard course of IMRT has been given. In addition, the investigators will look at whether magnetic resonance imaging (MRI) scanning can detect treatment response in oropharynx tumors earlier than with standard tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age with histologically proven squamous cell carcinoma of the oropharynx
* HPV-negative disease status by routine p16 immunohistochemical (IHC) staining or in situ hybridization (ISH) of biopsied tumor tissue or >10 pack-year cigarette smoking history
* Stage T1-4, N0-3 disease, as defined by American Joint Committee on Cancer (AJCC) criteria
* Eastern Cooperative Oncology Group (ECOG) (Zubrod) Performance Status 0-2.

Exclusion Criteria:

* Patients who have undergone resection of primary disease
* Patients who have received induction chemotherapy for their oropharynx cancer diagnosis
* Prior cancer diagnosis within 5 years, except appropriately treated localized epithelial skin cancer or cervical cancer
* Prior radiation therapy to the head and neck region
* Women of childbearing potential (a woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 months]) and male participants must practice effective contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study
* Patient unable to tolerate MRI or having an estimated Glomerular Filtration Rate (GFR) <60 ml/min/1.73 m2.
* Severe, active co-morbidity, defined as follows:
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
* Transmural myocardial infarction within the last 6 months
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
* Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients
* History or treatment with potent immunosuppressive drugs for such conditions as organ transplant, severe rheumatoid arthritis, etc. within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Safety and dose-limiting toxicity of dose escalated stereotactic radiotherapy in patients with high-risk oropharyngeal squamous cancer using (CTCAE), version 4.03 | up to two years post SRS Boost
  study completed.

SECONDARY OUTCOMES:
Disease response using Revised RECIST guideline (version 1.1) | up to two years post SRS Boost
  study completed

CONTACTS AND LOCATIONS:
Overall Officials: Maged Ghaly, MD, Principal Investigator — Northwell Health- Center for Advanced Medicine
Locations (1):
- Northwell Health- Center for Advanced Medicine, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vempati P, Halthore AN, Teckie S, Rana Z, Gogineni E, Antone J, Zhang H, Marrero M, Beadle K, Frank DK, Aziz M, Paul D, Ghaly M. Phase I trial of dose-escalated stereotactic radiosurgery (SRS) boost for unfavorable locally advanced oropharyngeal cancer. Radiat Oncol. 2020 Dec 11;15(1):278. doi: 10.1186/s13014-020-01718-w. PMID 33308265